CLINICAL TRIAL: NCT03151824
Title: Gender-specific Associations Between Quality of Life and Leukocyte Telomere Length: A Cross-sectional Study
Brief Title: Gender-specific Associations Between Quality of Life and Leukocyte Telomere Length
Status: Completed | Type: Observational
Sponsor: Jung-Ha Kim (Other)
Responsible Party: Sponsor-Investigator, Jung-Ha Kim, Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Organization: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Other Study IDs: C 2013152(1112)
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Apparently Healthy People Aged 55 and Over
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: quality of life — Quality of life which was measured by the Korean version of the 36-item short-form health survey (SF-36)

SUMMARY:
Quality of life (QoL) is an important factor for successful aging. Telomere length is an indicator of cellular aging and cumulative biological stress and is thus related to health status and survival. However, the relationship between QoL and telomere length has not yet been examined. In this study we investigated the relationship between leukocyte telomere length (LTL) and QoL.

However, the relationship between overall QoL and LTL has not previously been investigated. Therefore, this study was conducted to examine the relationship between LTL and QoL. QoL was measured by the Korean version of the 36-item short-form health survey (SF-36), which is a multidimensional scale consisting of subjective evaluation.

ELIGIBILITY:
Inclusion Criteria:

* married couple
* apparently healthy subjects above 55 years

Exclusion Criteria:

* Subjects who had experienced hormone therapy
* Subjects who had been diagnosed with dementia, Parkinson's disease, stroke, ischemic heart disease, congestive heart failure, arrhythmia, depression, cancer, thyroid disorders, or chronic renal disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 164 apparently healthy subjects (82 couples) aged 55 and over were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2013-10-25 (Actual); Primary Completion 2014-10-24 (Actual); Study Completion 2014-10-24 (Actual)

PRIMARY OUTCOMES:
leukocyte telomere length | 8months
  Leukocyte telomere length was measured as telomere repeat copy number relative to single gene copy number by quantitative real-time PCR